CLINICAL TRIAL: NCT00301522
Title: TAXUS V: De Novo Lesion: A Randomized, Double-blind Trial to Assess TAXUS Paclitaxel-Eluting Coronary Stents, SR Formulation, in the Treatment of De Novo Coronary Lesions
Brief Title: Randomized Trial Evaluating Slow-Release Formulation TAXUS Paclitaxel-Eluting Coronary Stents to Treat De Novo Coronary Lesions
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Marcie Clarkin, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAXUS V De novo; S5442
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Stenosis
Keywords: Coronary; Artery; Stenosis; Drug-eluting; stent; restenosis; revascularization
MeSH Terms: conditions — Coronary Stenosis; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Paclitaxel-Eluting Coronary Stent, Slow-Formulation
- Arm 2 (Active Comparator)
  Interventions: Device: Express2

INTERVENTIONS:
Device: TAXUS Paclitaxel-Eluting Coronary Stent, Slow-Formulation — Paclitaxel-Eluting Coronary Stent, Slow-Formulation
  Arms: Arm 1
Device: Express2 — Coronary Stent System
  Arms: Arm 2

SUMMARY:
The primary objective of this study is to further evaluate the safety and effectiveness of the TAXUS Express2 Paclitaxel-Eluting Coronary Stent System in long lesion lengths, small and large vessel diameters and with multiple overlapping stents in the treatment of de novo coronary artery lesions

DETAILED DESCRIPTION:
The primary endpoint is the incidence rate of TVR through 9 months post index procedure. In this protocol, TVR must be ischemia driven, based on the presence of symptoms, positive functional testing or Quantitative Coronary Angiography (QCA) severity of restenosis.

Secondary endpoints include the following:

* Incidence rates of composite MACE and the individual components of MACE assessed at discharge, 1, 4 and 9 months post index procedure and annually for 5 years (i.e., 1, 2, 3, 4 and 5 years post index procedure).
* Stent thrombosis rate.
* TVF.
* Clinical procedural success and technical success.
* Binary restenosis rate.
* Additional angiographic endpoints to be measured in all patients with 9 month angiographic follow-up include:

  * Absolute lesion length
  * Reference Vessel Diameter (RVD)
  * Minimum Lumen Diameter (MLD)
  * Percent diameter stenosis (% DS)
  * Acute gain
  * Late loss
  * Loss index
  * Patterns of recurrent restenosis, including edge effect
  * Coronary aneurysm
* IVUS Substudy

  * Identification of potential safety issues, i.e., incomplete stent apposition.
  * change in neointimal volume from post procedure to follow-up
  * change in MLD within stent
  * minimum lumen area (MLA) within stent
  * lumen, plaque and vessel measurements at the stent edges (outside stent)

ELIGIBILITY:
Inclusion Criteria:

* Patient was ≥ 18 years old.
* Eligible for percutaneous coronary intervention.
* Documented stable angina pectoris.
* LVEF of greater than 25%.
* Acceptable candidate for coronary artery bypass grafting.
* Target lesion segment is located within a single native coronary vessel.
* Target lesion was de novo.
* RVD was greater than 2.25 mm and less than 4.0 mm .and patient and/or lesion fulfilled protocol defined subgroups.
* Cumulative target lesion length was greater than 10 mm and less than 46mm assessed after pre-dilatation with standard balloon or cutting balloon angioplasty, including adjacent areas of dissection that were covered.
* Target lesion diameter stenosis less than 50% before pre-dilatation .
* Vessel and lesion morphology such that the lesion was treated only with study stent(s); no planned use of commercial stents.

Exclusion Criteria:

* Known hypersensitivity to paclitaxel.
* Any previous or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent.
* Planned use of both the study stent and a non-study stent in the treatment of the target vessel.
* Previous or planned treatment with intravascular brachytherapy in the target vessel.
* Recent MI.
* CK-MB greater than 2x the local laboratory's upper limit of normal.
* Cerebrovascular accident within 6 months of randomization.
* Planned CABG ≤ 9 months post index procedure.
* Acute or chronic renal dysfunction.
* Leukopenia.
* Thrombocytopenia or thrombocytosis.
* Active peptic ulcer or active gastrointestinal bleeding, or previously active within 6 months.
* Known allergy to stainless steel.
* Any prior true anaphylactic reaction to contrast agents.
* Contraindication to ASA or to both clopidogrel and ticlopidine.
* Patient was on warfarin or it was anticipated that treatment with warfarin would have been required during any period within 6 months post the index procedure.
* Patient was or had been treated with chemotherapeutic agents within 12 months of the index procedure.
* Anticipated treatment with paclitaxel, oral rapamycin or colchicine during any period in the 9 months post index procedure.
* Male or female with known intention to procreate within 3 months post index procedure.
* Co-morbid condition(s) that could limit the patient's ability to participate in the study, limit compliance with follow-up requirements or impact the scientific integrity of the study.
* Planned surgical procedure requiring withdrawal of any anti-platelet therapy within 6 months post index procedure.
* Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.
* Unprotected left main coronary artery disease.
* Target lesion was ostial in location.
* Target lesion and/or target vessel proximal to the target lesion was moderately or severely calcified.
* Target lesion was located within or distal to a > 60° bend in the vessel.
* Side branch of the target lesion included ostial narrowing ≥ 50% DS and was ≥ 2.0 mm diameter.
* Target lesion was totally occluded.
* Angiographic presence of probable or definite thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2003-02; Primary Completion 2004-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence rate of TVR through 9 months post index procedure | 9 Months

SECONDARY OUTCOMES:
• Incidence rates of composite MACE and the individual components of MACE assessed at discharge, 1, 4 and 9 months post index procedure and annually for 5 years (i.e., 1, 2, 3, 4 and 5 years post index procedure). | 5 Years
Stent thrombosis rate | 5 Years
Target Vessel Failure | 5 Years
Clinical procedural success and technical success | 5 years
Binary restenosis rate. | 5 Years
Absolute lesion length | 9 Months
Reference Vessel Diameter (RVD) | 9 Months
Minimum Lumen Diameter (MLD) | 9 Months
Percent diameter stenosis (% DS) | 9 Months
Acute gain | 9 Months
Late loss | 9 Months
Loss index | 9 Months
Patterns of recurrent restenosis, including edge effect | 9 Months
Coronary aneurysm | 9 Months
Identification of potential safety issues, i.e., incomplete stent apposition. | 9 Months
change in neointimal volume from post procedure to follow-up | 9 Months
change in MLD within stent | 9 Months
minimum lumen area (MLA) within stent | 9 Months
lumen, plaque and vessel measurements at the stent edges (outside stent) | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, MD, Principal Investigator — Columbia University; Stephen G. Ellis, MD, Principal Investigator — The Cleveland Clinic
Locations (72):
- United States (72):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Cardiovascular Associates PC/Baptist Medical Center Montclair, Birmingham, Alabama
  - UAB Interventional Cardiology, Birmingham, Alabama
  - Arizona Heart Institute and Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital LaJolla, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Stanford Medical Center, Stanford, California
  - Aurora Denver Cardiology, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Heart Research Institute, LLC, Atlantis, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Miami International Cardiology Consultants, Miami Beach, Florida
  - Mediquest Research Group, Inc., Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - The Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic/Saint Mary's Hospital, Rochester, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Albany Medical Center/Capital Cardiovascular Associates, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Mid-Carolina Cardiology Research Division/Presbyterian Hospital, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MidWest Cardiology Research Foundation/Riverside Methodist Hospital, Columbus, Ohio
  - North Ohio Research, Ltd, Elyria, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - St. Mary's Medical Center, Langhorne, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - South Carolina Heart Center, Columbia, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
  - South Austin Hospital/Capital Cardiovascular Specialists, Austin, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Houston Hermann Hospital, Houston, Texas
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Stone GW, Ellis SG, Cannon L, Mann JT, Greenberg JD, Spriggs D, O'Shaughnessy CD, DeMaio S, Hall P, Popma JJ, Koglin J, Russell ME; TAXUS V Investigators. Comparison of a polymer-based paclitaxel-eluting stent with a bare metal stent in patients with complex coronary artery disease: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1215-23. doi: 10.1001/jama.294.10.1215. PMID 16160130
- [Derived] Wakabayashi K, Mintz GS, Weissman NJ, Stone GW, Ellis SG, Grube E, Ormiston JA, Turco MA, Pakala R, Xue Z, Desale S, Laynez-Carnicero A, Romaguera R, Sardi G, Pichard AD, Waksman R. Impact of drug-eluting stents on distal vessels. Circ Cardiovasc Interv. 2012 Apr;5(2):211-9. doi: 10.1161/CIRCINTERVENTIONS.111.965780. Epub 2012 Apr 10. PMID 22496083
- [Derived] Doi H, Maehara A, Mintz GS, Yu A, Wang H, Mandinov L, Popma JJ, Ellis SG, Grube E, Dawkins KD, Weissman NJ, Turco MA, Ormiston JA, Stone GW. Impact of post-intervention minimal stent area on 9-month follow-up patency of paclitaxel-eluting stents: an integrated intravascular ultrasound analysis from the TAXUS IV, V, and VI and TAXUS ATLAS Workhorse, Long Lesion, and Direct Stent Trials. JACC Cardiovasc Interv. 2009 Dec;2(12):1269-75. doi: 10.1016/j.jcin.2009.10.005. PMID 20129555